CLINICAL TRIAL: NCT03692104
Title: Comparison Between Postoperative Ultrasound-CT Fusion With MRI-CT Fusion for Postimplant Dosimetry for Prostate LDR Permanent Seed Brachytherapy
Brief Title: US-CT Fusion for Post Implant Dosimetry
Status: Completed | Type: Observational
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Juanita Crook, Radiation Oncologist, British Columbia Cancer Agency
Other Study IDs: H17-02634
Record Dates: First submitted 2018-09-27; First posted 2018-10-02 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; brachytherapy; Quality assurance
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: transrectal ultrasound — Use of US for post implant quality assessment

SUMMARY:
Post implant dosimetry is an essential part of quality assurance after permanent seed prostate brachytherapy. CT imaging is the standard of assessment but due to contouring uncertainties, MR-CT fusion is preferred. This is not always available due to financial restrictions. This study explores the possibility of post implant US-CT fusion to improve contouring accuracy and potentially replace the use of MR-CT fusion.

DETAILED DESCRIPTION:
25 participants undergoing permanent seed prostate brachytherapy will be approached to undergo collection of prostate US images at the completion of their procedure. This will add approximately 5 minutes to the duration of their brachytherapy procedure. The US study will not entail any discomfort or risk to participants as they are still under anesthesia for the implant procedure. The institution standard of care for quality assurance will be complied with, obtaining a CT and MRI of the prostate at 30 days after the procedure. These will be co-registered and analyzed in the normal fashion. In addition, the post implant US images will also be co-registered with the CT and the resulting dosimetric parameters compared.

ELIGIBILITY:
Inclusion Criteria:

* localized prostate cancer suitable for permanent seed implant brachytherapy as either monotherapy or as a boost

Exclusion Criteria:

* Unable to undergo MRI

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing prostate brachytherapy for localized prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of prostate dosimetry assessed by US-CT fusion with respect to the standard MR-CT fusion | 1 month
  Dosimetry will be calculated using 2 different imaging modalities (US vs MRI) and compared

SECONDARY OUTCOMES:
Comparison of prostate volume assessed by 2 different imaging modalities | 1 month
  Assessment of prostate volume as contoured on US vs MRI post implant

CONTACTS AND LOCATIONS:
Overall Officials: Francois Bachand, MD, Study Chair — BC Cancer
Locations (1):
- BC Cancer, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No